CLINICAL TRIAL: NCT05774158
Title: Investigation of Adults With Congenital Heart Disease in the Scope of the International Classification of Functioning, Disability, and Health
Brief Title: Investigation of Adults With Congenital Heart Disease in the Scope of the ICF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Tuğba Siyah, Principal Investigator, Hacettepe University
Other Study IDs: 03032023
Record Dates: First submitted 2023-03-07; First posted 2023-03-17 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2023-03

CONDITIONS: Congenital Heart Disease; ICF; Quality of Life
Keywords: congenital heart disease; ICF; muscle strength; physical activity; quality of life
MeSH Terms: conditions — Heart Defects, Congenital; Motor Activity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult Congenital Heart Diseases
  Interventions: Other: Physiotherapy assessment

INTERVENTIONS:
Other: Physiotherapy assessment — Of the individuals included in the study; Information about age, height, body weight, type of congenital heart disease, surgical history, drug use, comorbid chronic disease, education level and occupation will be obtained. Functional Capacity, Peripheral Muscular Strength, Hand Grip Strength, Fatigue, Physical Activity Level, Quality of Life, Social Participation, Depression Anxiety Stress Level and Physical Activity Barriers will be evaluated

SUMMARY:
Congenital heart disease (CHD) is one of the common birth defects with a prevalence of approximately 1 in 1000 live births worldwide. While 15% of patients with CHD reached adulthood in the past, this rate is close to 90% today thanks to advancing medicine and technology.As individuals with CHD age, they may be affected by acquired cardiovascular risk factors common in the general population in addition to heart diseases such as arterial hypertension, obesity, and diabetes, increasing the risk of metabolic disease, stroke, and coronary artery disease. In addition to these risk factors, the disease affects both the social and familial environment of the patients. In addition to the mortality and morbidity of patients, which was the most important outcome measure in the past, quality of life has become the subject of current research. The International Classification of Functioning and Health (ICF) was adopted in 2001 for the use of a common, standard language and framework for describing health and health-related conditions, and is an international and standardized classification system that can evaluate functioning, disability and health holistically. There are no studies in the literature evaluating body structure, function and activity and participation in adults with congenital heart disease within the scope of ICF. Therefore, the aim of this study is; It is the evaluation of adults with CHD according to ICF sub-parameters (body structure and functions, activity and participation, and environmental factors) and the correlation of ICF parameters with other evaluation methods.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with congenital heart disease
* Being between the ages of 18-65
* To have been informed about the study and given written consent to participate in the study.

Exclusion Criteria:

* Having a neurological, orthopedic or any systemic disease,
* Presence of infection and malignancy,
* Cognitive, psychological and mental status are not suitable for evaluations,
* To undergo another surgery other than cardiac surgery.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults with congenital heart disease
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-08-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
6-minute walking test | December 2022- August 2023
  Functional capacities of individuals will be evaluated with the 6-minute walking test (6MWT). With the 6MWT, it provides the evaluation of the functional capacities of the cardiac, respiratory and neuromuscular systems of the participants and the evaluation of the responses to exercise. For 6MWT, the start and end places of a 30-meter area will be marked, and the patients will be asked to walk this distance for 6 minutes without running at the maximum walking speed they can walk. After 6 minutes, the distance walked will be recorded in meters.
Peripheral Muscle Strength | December 2022- August 2023
  Knee extensor and shoulder abductor muscle strength will be evaluated with a digital dynamometer (Lafayette, USA). Muscle strength measurements will be applied from both the right and left side extremities of the participant in triplicate and the average of the values will be recorded in kilopascals.
Hand Grip Strength | December 2022- August 2023
  Maximum isometric hand grip strength will be evaluated with the electronic hand dynamometer Jamar (Performance Health; United States). Three separate measurements will be made for the right and left hands, and the average of the measurements will be recorded in kilopascals. A 20-second rest period will be given between measurements. During the evaluation, the evaluation will be made while the patient is in a sitting position with back support.
Evaluation of Fatigue | December 2022- August 2023
  The effect of the fatigue levels of the participants on the functions will be evaluated with the Fatigue Severity Scale. In this scale, the participants are asked to give points between 1-7 for the questions asked considering their last week. The total score is calculated by dividing the total score by the number of questions. A score of 4 or higher usually indicates severe fatigue.
Physical Activity Level | December 2022- August 2023
  The International Physical Activity Questionnaire (IPAQ) will be used to assess the physical activity level of the participants. The International Physical Activity Questionnaire (IPAQ) is a standard tool for measuring physical activity, developed by researchers from various countries with support from the World Health Organization and the Centers for Disease Control. The questionnaire is filled in the last 7 days, taking into account the physical activity level of the participants. According to the total physical activity score, the physical activity levels of the participants are classified as low, medium and high.
Measurement of quality of life | December 2022- August 2023
  The quality of life of the participants will be evaluated with the Multidimensional Quality of Life Scale. The scale is a 35-item scale that covers nine sub-dimensions and each sub-dimension includes 4 items. The answers in the scale are numbered from 1 to 7. 1 is expressed as "not at all satisfied" and "7" is expressed as "very satisfied". The sub-dimensions of the questionnaire; mental health, physical health, physical function, cognitive function, sexual function, social function, productivity, access to health personnel and financial situation.
Evaluation of Participation | December 2022- August 2023
  The revised form of the Community Participation Questionnaire (TKA-R) will be used to assess participation in the study. TKA-R consists of 4 sub-units as home participation, social participation, productivity, electronic social network and a total of 18 questions. Scoring focuses primarily on the frequency of performing the activity or social role, and secondly, on whether he/she does the activity alone or with family members. Questions are mostly evaluated between "0" and "2" points. The 2 points that can be taken from the questions represent a higher level of independence and social participation. The highest score that can be obtained from the survey is 35.
Depression Anxiety Stress | December 2022- August 2023
  The 21-item short form of the Depression, Stress and Anxiety Scale will be used to measure the depression, anxiety and stress levels of the participants. There are 7 questions in each scale to measure the dimensions of depression, stress and anxiety. The scale is a 4-point Likert Type Scale; 0 "not suitable for me", 1 "somewhat suitable for me", 2 "usually suitable for me", and 3 "completely suitable for me". An increase in the scale score indicates an increase in the level of depression, stress and anxiety.
Physical Activity Barriers | December 2022- August 2023
  The Physical Activity Disability Scale for Adults will be used to identify the factors causing physical activity limitation of the participants. The Turkish version of the scale consists of 22 items. Personal barriers that cause physical activity limitation, social environment and physical environment are scored. Higher scores indicate the magnitude of barriers to physical activity.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No